CLINICAL TRIAL: NCT06201923
Title: The Efficacy of Thyme Honey Mouth Rinse on Polypharmacy-induced Xerostomia (A Randomized Controlled Clinical Trial With a Biochemical Assessment)
Brief Title: The Efficacy of Thyme Honey Mouth Rinse on Polypharmacy-induced Xerostomia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Neven Nabil Tadry Banoud, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Thyme Honey Mouth Rinse
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-01

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 0.2% thyme honey mouth rinse as intervention
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Thyme H) (Experimental): 0.2% thyme honey mouth rinse (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day.
  Interventions: Drug: Honey Mouthwash
- Group II (Saline G) (Placebo Comparator): normal saline oral rinse
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Honey Mouthwash — 0.2% thyme honey mouth rinse
  Other Names: thyme honey mouth rinse
  Arms: Group I (Thyme H)
Drug: Normal saline — 0.9% sodium chloride
  Other Names: saline mouth rinse
  Arms: Group II (Saline G)

SUMMARY:
The study is designed to evaluate the clinical efficacy of thyme honey as a mouth rinse in the management of polypharmacy-induced xerostomia concerning the unstimulated whole salivary flow rate and quality of life of patients along with a biochemical assessment of salivary nitric oxide levels.

DETAILED DESCRIPTION:
Saliva is a vital component in the mouth and the preservation of humans' general health depends on good oral health. Saliva contains primarily water (99.5%), followed by a 0.3% mixture of inorganic salts, enzymes, and proteins. There are many functions of saliva such as lubrication, microbial homeostasis, tooth protection, digestion process, taste, buffering, mineralization, and wound healing. So, when the salivary flow or composition changes due to various causes, these functions will be lost. The normal unstimulated salivary flow rate is about 0.3-0.4 ml/min, whereas the stimulated rate is 1.5-2.0 ml/ min. When there is an objective hyposalivation (< 0.1- 0.2 ml/min unstimulated or < 0.5 - 0.7 ml/min stimulated), patients frequently complain of xerostomia. Xerostomia can be defined as a subjective feeling of oral dryness that might be associated with a real decline in the salivary flow. It can be considered a major problem that greatly affects a person's quality of life due to dysphagia occurrence and taste sensation impairment. The prevalence of xerostomia in the general population ranged from 0.9% to 46%. So, it constitutes a serious health issue requiring attention. The causes of xerostomia can be categorized as systemic or local, depending on their nature. Furthermore, xerostomia is classified as permanent or periodic based on how long the symptoms last. Systemic causes of xerostomia included endocrinological (e.g., diabetes mellitus, autoimmune thyroid diseases), autoimmune (e.g., Sjogren's syndrome, rheumatoid arthritis, systemic lupus erythematosus), infectious (e.g., hepatitis C virus), and granulomatous (e.g., tuberculosis and sarcoidosis) diseases, while Local factors of xerostomia comprised multiple medications (polypharmacy), radical radiotherapy for the treatment of head and neck malignancies, and lifestyle factors, such as alcohol, tobacco, and caffeine consumption. Recently, it was also documented that 45.9% of patients with confirmed SARS-CoV-2 infection experienced xerostomia, with a considerable majority (76.5%) of them noting that it was their first time experiencing xerostomia. Polypharmacy is thought to be the most common cause of xerostomia. Several definitions of polypharmacy were reported in the literature. There was a wide range of numerical-only definitions of polypharmacy, ranging from two or more medications to 11 or more medications, Also the numerical definitions of polypharmacy incorporating duration of therapy ranged from the use of two or more medications for more than 240 days (long-term use) to five to nine medications used for 90 days or more, While descriptive definitions explained co-prescribing multiple medications and simultaneous and long-term use of different drugs by the same individual. More than 400 drugs have an impact on the function of the salivary glands and promote the development of xerostomia. Drugs that frequently contribute to xerostomia include antiparkinsonian pharmaceuticals, antipsychotics, antidepressants, anticholinergic, antihistamines, tranquilizers, oral hypoglycemics, diuretics, opioids, cytotoxic agents, and antihypertensive medications. The precise processes by which some drugs produce xerostomia aren't yet understood.

Various treatment modalities can be used to treat xerostomia and salivary hypofunction depending on the underlying cause of the condition, which are classified into systemic and topical agents. The FDA has approved systemic sialogogues, namely pilocarpine, and cevimeline, as a treatment modality. Cevimeline and the other medications are parasympathomimetics and act on muscarinic receptors. Despite their powerful effect, severe highly prevalent side effects are caused after their regular administration including vasodilatation, emesis, excessive sweating, hypotension, bronchoconstriction, increased urinary frequency, bradycardia, and vision problems. Topical and local medications for xerostomia continue to be a more appealing and secure therapy choice. These include sugar-free chewing gums, salivary stimulants, and substitutes. salivary substitutes make an effort to resemble natural saliva and act as oral lubricants without changing the salivary flow rate, and due to their viscosity, they are not commonly used and not accepted by most patients. These substitutes are mainly utilized when completely damaged salivary glands. Topical salivary stimulants are the most popular and widely tolerated among patients mainly used when there is residual functional salivary tissue. These topical stimulants can be divided into acid or mechanically-driven. Mechanical salivary stimulation occurs through the utilization of sugar-free chewing gums which aim to stimulate the major salivary glands to increase the salivary flow. While acid-driven stimulation occurs through acidification of the oral cavity with malic acid, and citric acid to increase the salivary flow rate. One of the topical salivary stimulants that have been recently studied is the thyme honey mouth rinse. Thyme honey is used for xerostomia under the assumption that it has saliva-stimulating effects as it consists of various organic acids such as ascorbic acid, citric acid, and malic acid which are used as saliva stimulators. Previous research has demonstrated that organic acids stimulate the chemoreceptors in the oral cavity, increasing the flow of saliva. Later, thyme honey has proven its efficacy in preventing radiation-induced salivary gland destruction and xerostomia. Thyme honey has antibacterial, antiviral, antifungal, anti-inflammatory, antioxidant, and anticarcinogenic properties. It has been used to treat burns, surgical wounds, and oral infections due to its antibacterial and analgesic properties and ability to promote epithelialization. The majority of honey varieties produce hydrogen peroxide when diluted due to the activation of the enzyme glucose oxidase, which oxidizes glucose to gluconic acid and hydrogen peroxide. The main component of honey's antibacterial activity is hydrogen peroxide as well as the presence of phytochemicals and its acidic environment with a pH ranging from 3.2 to 4.5.

Nitric oxide in the saliva is produced by the nerve ending in the salivary gland's endothelium and macrophages in response to the oral bacteria. Nitric oxide levels rise and oxidative stress occurs as a result of phagocyte induction. So, High levels of nitrate and nitrite (the stable end products of nitric oxide) in typical saliva help to locally produce nitrogen intermediates with possible antibacterial capabilities, enhanced mucosal blood flow, and improved oral mucus formation. The salivary NO level in patients with xerostomia is significantly lower than in those without xerostomia. So, salivary nitric oxide level could be considered a predictor of xerostomia.

A. Clinical Assessment: all patients are evaluated at baseline, 2 and 4 weeks after intervention through

1. Measurement of Unstimulated Salivary Flow Rate (UFR): by spitting method for assessment of salivary gland hypofunction. Measurements are expressed in millimeters per minute (ml/min). If the unstimulated flow rate is less than 0.2 mL/min. it will be considered to represent salivary gland hypofunction and this patient will be included in the study.
2. Measurement of subjective symptoms of oral dryness: by using a questionnaire consisting of four questions that assess the severity of dry mouth. patients will answer these questions with (yes or no). positive response to any question indicates a reduced unstimulated salivary flow rate and this patient will be included in the study.

   Q1: Does it seem like there isn't enough saliva in your mouth? Q2: Do you ever have trouble swallowing? Q3: Does eating a meal cause your mouth to feel dry? Q4: Do you drink liquids to make it easier to swallow dry food?
3. Measurement of objective signs of oral dryness: by using a clinical oral dryness score (CODS) consisting of a 10-point scale, each point representing a feature of dryness in the mouth. The clinician scores the features observed in the patient's mouth from 0-10. Patients with a score less than 2 will be excluded.

1. The buccal mucosa becomes stuck with the mirror. 2. The tongue adheres to the mirror. 3. Saliva with foam. 4. There isn't any saliva collecting on the mouth's floor. 5. The papillae of the tongue have disappeared. 6. Modified or smooth gingival structure. 7. The mucosa of the mouth, particularly the palate, appears glassy. 8. Lobular or fissured tongue. 9. Cervical caries that have just been repaired within the past six months (more than two teeth). 10. Debris on the palate (excluding under dentures).

All patients are also evaluated at baseline and after one month from intervention through the following:

4) Xerostomia-related quality of life questionnaire: includes 15 questions regarding how dry mouth affects a person's quality of life. The questions are:

1. Is the type or quantity of food you can eat restricted by your mouth dryness? 2. Does having a dry mouth make you uncomfortable? 3. Does your oral dryness make you anxious or concerned a lot? 4. Do you avoid social situations because of dry mouth? 5. Is it unsettling to eat in front of others when your mouth is dry? 6. When speaking in front of other people, does your dry mouth make you feel uneasy? 7. Does your oral dryness make you nervous? 8. Are you worried about how your teeth and mouth seem because of your mouth dryness? 9. Do you find it difficult to enjoy life because of your dry mouth? 10. Does having a dry mouth affect your everyday activities? 11. Does your mouth dryness affect the intimacy with your relationships? 12. Does dry mouth affect how well you can taste food? 13. Does having a dry mouth lessen your overall enjoyment of life? 14. Does your mouth dryness interfere with every part of your life? 15. How would you feel if you were forced to live the remainder of your days with a dry mouth the way it is right now? The questionnaire will be translated verbally, and answers will be collected orally from the patients and documented by an investigator not involved in assigning the intervention to patients.

B. Biochemical Assessment:

> Measurement of salivary nitric oxide (NO) level: measured at baseline and after one month in the Lab.

Statistical Methods:

All the data will be collected and analyzed statistically. Categorical data will be represented as frequency (n) and percentage (%) and will be analyzed using the chi-square test. Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values, and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was found to be normally distributed, it will be presented as mean and standard deviation values and an independent t-test will be used for the analysis. If the assumption of normality is found to be violated; the data will be presented as median and range values and will be analyzed using the Mann-Whitney U test. The significance level will be set at p ≤0.05 for all tests. Statistical analysis will be performed with IBM® SPSS® Statistics Version 26 for Windows.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders, aged between 40 and 65 years old.
2. Patients using two or more medications known to cause xerostomia or salivary hypofunction (e.g., anxiolytics, anorexiants, anti-asthmatics, anticholinergics, anti-depressants, anti-emetics, anti-histamines, antihypertensives, anti-parkinsonians, anti-psychotics, antithrombotics, muscle relaxants, anticonvulsants, decongestants, diuretics, NSAIDs, or sedatives). Patients taking previous drugs for 240 days or more before the start of the trial and expected to continue.
3. Patients are willing to follow all the instructions and attend all the study-associated visits.

Exclusion Criteria:

1. Patients who had received radiation therapy to the head and neck region.
2. Patients with other systemic diseases known to cause xerostomia (diabetes mellitus, Sjogren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, hepatitis C virus, tuberculosis, or sarcoidosis).
3. Patients using any other medication for their dry mouth condition (pilocarpine, cevimeline) 7 days before entering into the study.
4. Patients requiring hospitalization for any medical problem during the study.
5. Known hypersensitivity to the active ingredient of the product that will be used as assessed by the medical history questionnaire.
6. Vulnerable groups such as pregnant females, prisoners, and mentally or physically handicapped individuals.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the clinical efficacy of 0.2% thyme honey mouth rinse on salivary flow rate of patients having polypharmacy-induced xerostomia | one month
  To eliminate any circadian changes, the unstimulated salivary flow rate will be measured for all patients between 9:00 to 11:00 a.m. Before saliva collection, participants are requested to wait at least two hours without eating, drinking, or brushing their teeth. Then, after swallowing all the saliva present in their mouth, unstimulated whole saliva will be collected by spitting method every 60s for 5 min in a sterile tube. The tubes are kept in a refrigerator (-20 centigrade) before sending them to the laboratory to prevent changing the composition of the saliva.

SECONDARY OUTCOMES:
Evaluate the clinical effect of thyme honey mouth rinse on the quality of life of the patients as well as its biochemical effect on the level of salivary nitric oxide | one month
  Xerostomia-related quality of life questionnaire which includes 15 questions will be used.
  salivary nitric oxide level will be assessed by Nitric Oxide Assay Kit (Colorimetric) based on the Griess reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan S. Ibrahim, Prof., Study Director — Professor of Oral Medicine, Periodontology, Faculty of Dentistry, Ain Shams University; Ola M. Ezzatt Hassanein, Ass. Prof., Study Director — Associate Professor of Oral Medicine, Periodontology, Faculty of Dentistry, Ain Shams University
Locations (1):
- Faculty of dentistry Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humphrey SP, Williamson RT. A review of saliva: normal composition, flow, and function. J Prosthet Dent. 2001 Feb;85(2):162-9. doi: 10.1067/mpr.2001.113778. PMID 11208206
- [Background] Cassolato SF, Turnbull RS. Xerostomia: clinical aspects and treatment. Gerodontology. 2003 Dec;20(2):64-77. doi: 10.1111/j.1741-2358.2003.00064.x. PMID 14697016
- [Background] Pedersen AM, Bardow A, Jensen SB, Nauntofte B. Saliva and gastrointestinal functions of taste, mastication, swallowing and digestion. Oral Dis. 2002 May;8(3):117-29. doi: 10.1034/j.1601-0825.2002.02851.x. PMID 12108756
- [Background] Napenas JJ, Brennan MT, Fox PC. Diagnosis and treatment of xerostomia (dry mouth). Odontology. 2009 Jul;97(2):76-83. doi: 10.1007/s10266-008-0099-7. Epub 2009 Jul 29. PMID 19639449
- [Background] Masnoon N, Shakib S, Kalisch-Ellett L, Caughey GE. What is polypharmacy? A systematic review of definitions. BMC Geriatr. 2017 Oct 10;17(1):230. doi: 10.1186/s12877-017-0621-2. PMID 29017448
- [Background] Barbe AG. Medication-Induced Xerostomia and Hyposalivation in the Elderly: Culprits, Complications, and Management. Drugs Aging. 2018 Oct;35(10):877-885. doi: 10.1007/s40266-018-0588-5. PMID 30187289
- [Background] Charalambous A, Lambrinou E, Katodritis N, Vomvas D, Raftopoulos V, Georgiou M, Paikousis L, Charalambous M. The effectiveness of thyme honey for the management of treatment-induced xerostomia in head and neck cancer patients: A feasibility randomized control trial. Eur J Oncol Nurs. 2017 Apr;27:1-8. doi: 10.1016/j.ejon.2017.01.001. Epub 2017 Jan 16. PMID 28279391
- [Background] Charalambous M, Raftopoulos V, Paikousis L, Katodritis N, Lambrinou E, Vomvas D, Georgiou M, Charalambous A. The effect of the use of thyme honey in minimizing radiation - induced oral mucositis in head and neck cancer patients: A randomized controlled trial. Eur J Oncol Nurs. 2018 Jun;34:89-97. doi: 10.1016/j.ejon.2018.04.003. Epub 2018 Apr 30. PMID 29784145
- [Background] Biswal BM, Zakaria A, Ahmad NM. Topical application of honey in the management of radiation mucositis: a preliminary study. Support Care Cancer. 2003 Apr;11(4):242-8. doi: 10.1007/s00520-003-0443-y. Epub 2003 Feb 19. PMID 12673463
- [Background] Osailan SM, Pramanik R, Shirlaw P, Proctor GB, Challacombe SJ. Clinical assessment of oral dryness: development of a scoring system related to salivary flow and mucosal wetness. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Nov;114(5):597-603. doi: 10.1016/j.oooo.2012.05.009. Epub 2012 Sep 7. PMID 22959491
- [Background] Ship JA, McCutcheon JA, Spivakovsky S, Kerr AR. Safety and effectiveness of topical dry mouth products containing olive oil, betaine, and xylitol in reducing xerostomia for polypharmacy-induced dry mouth. J Oral Rehabil. 2007 Oct;34(10):724-32. doi: 10.1111/j.1365-2842.2006.01718.x. PMID 17824884
- [Background] Carpenter GH. The secretion, components, and properties of saliva. Annu Rev Food Sci Technol. 2013;4:267-76. doi: 10.1146/annurev-food-030212-182700. PMID 23464573
- [Background] Afsaneh Abadi P, Koopaie M, Montazeri R. Comparison of salivary nitric oxide and oral health in diabetic patients with and without xerostomia. Diabetes Metab Syndr. 2020 Jan-Feb;14(1):11-15. doi: 10.1016/j.dsx.2019.11.014. Epub 2019 Nov 25. PMID 31809967
- [Background] Jockel-Schneider Y, Schlagenhauf U, Stolzel P, Gossner S, Carle R, Ehmke B, Prior K, Hagenfeld D. Nitrate-rich diet alters the composition of the oral microbiota in periodontal recall patients. J Periodontol. 2021 Nov;92(11):1536-1545. doi: 10.1002/JPER.20-0778. Epub 2021 Apr 6. PMID 33742692
- See also: The identification of inhibine, the antibacterial factor in honey, as hydrogen peroxide and its origin in a honey glucose-oxidase system — http://linkinghub.elsevier.com/retrieve/pii/0006300263903597
- See also: Measuring salivary flow: Challenges and opportunities — http://linkinghub.elsevier.com/retrieve/pii/S0002817714638800
- See also: Subjective reports of xerostomia and objective measures of salivary gland performance — http://linkinghub.elsevier.com/retrieve/pii/S0002817787540120